CLINICAL TRIAL: NCT00923741
Title: An Open Label Pilot Study to Evaluate the Effect on the Immune System of Talactoferrin in Adults With Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Effect of Talactoferrin in Adults With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080166; 08-C-0166; NCT00709943 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2012-11-06

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Lung Cancer; Immunity; Clinical Response; Cytokines; Elispot Assay; Non-Small Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — talactoferrin alfa; Blood Component Removal

INTERVENTIONS:
Drug: Talactoferrin
Procedure: Apheresis

SUMMARY:
Background:

More effective therapies are needed for patients with non-small cell lung cancer (NSCLC) whose disease has advanced or spread beyond the original site following standard treatment.

Talactoferrin is a genetically engineered form of the human protein lactoferrin, found in body secretions such as breast milk, tears and saliva.

In previous studies, talactoferrin improved life span in patients with NSCLC without causing toxic side effects.

Objectives:

To examine the effects of talactoferrin on the immune system and determine its effectiveness in treating NSCLC.

Eligibility:

Patients with advanced NSCLC who have tissue type HLA-A2 and whose cancer has gotten worse following at least one course of treatment.

Design:

Talactoferrin treatment: Patients take liquid talactoferrin twice a day for 12 weeks, followed by 2 weeks off the drug. Treatment may continue in these 14-week cycles depending on the drug side effects and the response of the tumor.

Evaluations: Patients are evaluated at the clinic with a physical examination, check of vital signs and blood tests every 3 weeks.

CT scans: Patients have CT scans to monitor disease before starting treatment, again at 6 weeks and 12 weeks and then every 12 weeks during the duration of treatment.

Apheresis: Quantities of white blood cells called lymphocytes are collected through a procedure called apheresis in order to measure the immune response to treatment. In this procedure, blood is collected through a needle placed in a vein in the arm (similar to donating blood) and circulated through a cell separator machine. The lymphocytes are extracted and the rest of the blood is returned to the body through the same needle.

DETAILED DESCRIPTION:
Background:

Patients with locally advanced or metastatic NSCLC have a very poor prognosis even with surgery, chemotherapy, and radiation treatments.

Patients who respond to 1st line chemotherapy invariably develop disease progression, and their median survival is between 6-8 months.

Talactoferrin alfa (TLF) is a recombinant human lactoferrin.

TLF displays anti-infective (against bacteria, viruses, protozoa and fungi) and anti-inflammatory properties, anti-tumor activity and anti-asthma properties.

Preclinical studies have demonstrated an increase in cytokines that stimulate both innate and adaptive immunity, as well as increasing the numbers of NK-T cells and CD8+ T-lymphocytes found in Peyer s Patches.

Previous studies in NSCLC have demonstrated safety and evidence of clinical activity.

Objectives:

Primary: To evaluate the effects of administration of talactoferrin to patients with advanced non-small cell lung cancer on the quantitative and functional changes in CD4, CD8, NK, and Treg populations in peripheral blood mononuclear cells (PBMC) and on the levels of cytokines and chemokines in serum.

Secondary: To evaluate clinical response to talactoferrin. To evaluate the safety of talactoferrin.

Eligibility:

Patients with cytologically or histologically confirmed progressive, recurrent, or refractory stage IIIb or IV NSCLC.

Patients must be HLA-A2 positive.

Design:

Single-arm pilot study

Ten patients will be enrolled to receive daily oral talactoferrin (1.5 g/ bid) for up to 12 weeks.

Patients who benefit from treatment will be able to continue on a 12 weeks on 2 weeks off schedule until progression.

Evaluation will be performed every 3 weeks with CT chest, abdomen, and pelvis at baseline, week 6, and week 12.

Immunologic studies (including apheresis) will be performed at baseline, week 6, and week 12.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age greater than or equal to 18 years

Histologically or cytologically confirmed progressive, recurrent, or refractory stage IIIB or IV NSCLC; confirmation of pathologic diagnosis to be conducted at the NCI Laboratory of Pathology

Patients may not be eligible for other curative intent treatment (e.g., surgical resection). For the purpose of eligibility for this trial, the above-cited disease states are defined as follows:

* Progressive NSCLC defined as increasing measurable disease, or the appearance of new measurable disease by RECIST criteria.
* Recurrent NSCLC defined as the reappearance of measurable disease or the appearance of new measurable disease by RECIST criteria after prior successful treatment or complete response.
* Refractory NSCLC defined as achieving less than a complete response and having residual measurable disease by RECIST criteria after prior treatment with chemotherapy, targeted or small molecules, monoclonal antibodies, or any combination of these.
* Patients may enroll who are not candidates for, or who have documented refusal to receive standard therapy (e.g., chemotherapy) for their disease.

HLA-A2 allele

Patient must have evaluable or measurable disease

Total bilirubin less than or equal to 1.5 mg/dL (OR in patients with Gilbert s syndrome, a total bilirubin less than or equal to 3.0)

Creatinine less than 1.5 times Upper Limit of Normal (ULN) if greater than 1.5 times ULN, creatinine clearance on a 24 hour urine collection of greater than 60 mL/min.

AST (SGOT) and ALT (SGPT) less than or equal to 2.5 times the upper limit of normal (ULN); in case of liver metastases less than or equal to 5 x ULN

Eastern Cooperative Oncology Group (ECOG) score 0, 1, or 2

Able to understand and give informed consent

Recovered completely from any reversible toxicity associated with recent therapy. Typically this is 3-4 weeks for patients who most recently received cytotoxic therapy except for the nitrosoureas and mitomycin C for which 6 weeks is needed for recovery.

Hematological eligibility parameters (within 16 days of starting therapy):

* Granulocyte count greater than or equal to 1,500/mm(3)
* Platelet count greater than or equal to 75,000/mm(3)
* Hgb greater than or equal to 9 Gm/dL

EXCLUSION CRITERIA:

Presence of brain metastases, unless the patient received brain irradiation at least 4 weeks prior to enrollment, and is stable, asymptomatic, and off steroids for at least 4 weeks prior to registration

History of allergic reactions to compounds of similar chemical or biologic composition to Talactoferrin. At this point, no specific compounds have been identified.

History of other malignancies except: (i) adequately treated basal or squamous cell carcinoma of the skin; (ii) curatively treated, a) in situ carcinoma of the uterine cervix, b) prostate cancer, or c) superficial bladder cancer; or (iii) other curatively treated solid tumor with no evidence of disease for greater than or equal to 5 years

Uncontrolled ischemic heart disease, or uncontrolled symptomatic congestive heart failure

Serious active infection

Psychiatric illness/ social situations that would limit study compliance

Other uncontrolled serious chronic disease or conditions that in the investigator s opinion could render compliance or follow-up in the protocol problematic

Concurrent radiotherapy or radiotherapy within 4 weeks prior to enrollment or previous radiotherapy to the target lesion sites (the sites that are to be followed for determination of a response)

Concurrent use of topical steroids (including steroid eye drops) or systemic steroids. Nasal or inhaled steroid use is permitted.

HIV positive

Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease)

History of opportunistic infections

Hepatitis B surface antigen positive or hepatitis C positive

Receipt of any investigational medication within 4 weeks prior to enrollment.

Pregnant or lactating patients, or fertile female patients with a positive pregnancy test (serum beta-human chorionic gonadotropin [beta-hCG] at screening and at baseline), or fertile female patients unwilling to use adequate contraception (including condom use, birth control pills, or IUD) during treatment and 30 days after completion of treatment

Sexually active male patients unwilling to practice contraception (condom use) while participating on the study and up to 30 days after completion of treatment

Legal incapacity or limited legal capacity, unless authorization is granted by a legal guardian

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-06-19; Primary Completion 2010-02-01 (Actual); Study Completion 2010-02-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of talactoferrin to patients with advanced NSCLC on quantitative and functional changes in CD4, CD8, NK, and Treg populations in peripheral blood mononuclear cells (PBMC) and on the levels of cytokines and chemokines in s...

SECONDARY OUTCOMES:
To evaluate clinical response to talactoferrin. To evaluate the safety of talactoferrin.

CONTACTS AND LOCATIONS:
Overall Officials: James L Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States